CLINICAL TRIAL: NCT00153218
Title: An Observational Study of Current Practice Pattern on the Treatment of Women With Metastatic Breast Cancer Whose Tumors Overexpress Her2neu
Status: Completed | Type: Observational
Sponsor: Cancer Research Network (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: H2933s; CRN006
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: Metastatic Breast Cancer; Her2neu; trastuzumab
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to observe clinical outcomes of metastatic breast cancer patients whose tumors overexpress the Her2neu protein and are being treated with trastuzumab (Herceptin)either alone or combination with chemotherapy or hormonal therapy.

DETAILED DESCRIPTION:
In clinical practice, patients with metastatic breast cancer are being treated either with trastuzumab alone or trastuzumab in combination with chemotherapy or hormonal therapy as it has shown to increase survival. There is currently minimal information as to how long trastuzumab should be given after disease progresses on trastuzumab. This study is a chart review of the above-mentioned population which will capture information such as;

* what chemo or hormonal therapies are chosen by clinicians for Her-2 positive metastatic patients to combine with trastuzumab
* what the number of treatment regimens are (chemo or hormonal) given with trastuzumab
* what the clinical outcome of patients treated is
* what happens to the patients cardiac status with long term administration of trastuzumab
* what treatment patterns exist in the management of central nervous system metastases

This study aims to generate a hypotheses that can be tested from the information collected after is has been analyzed to give clinicians further meaningful data to guide treatment decisions beyond treatment progression.

ELIGIBILITY:
Inclusion Criteria:

* patients must have metastatic breast cancer
* tumor must have been determined to be Her-2 positive 3+ by immunohistochemistry or gene-amplified by fluorescence-in-situ hybridization (FISH)
* must have received trastuzumab alone or in combination with chemotherapy or hormonal therapy
* must not have received trastuzumab in the adjuvant or neoadjuvant setting
* must have started trastuzumab treatment for metastatic disease any time between January 1996 to June 2003

Exclusion Criteria:

* patients who received trastuzumab prior to 1996

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Her-2-neu positive breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Tan-Chiu, MD, Principal Investigator — Cancer Reserach Network, Inc.
Locations (2):
- United States (2):
  - Cancer Research Network, Inc., Plantation, Florida
  - University of Pittsburgh Cancer Institute Magee-Womans Hospital, Pittsburgh, Pennsylvania